CLINICAL TRIAL: NCT06597539
Title: A Prospective Study on Investigating the Value of 68Ga-grazytracer PET in Monitoring Responses to Immunotherapy of Advanced Hepatobiliary Malignancy
Brief Title: The Value of 68Ga-grazytracer PET in Monitoring Responses to Immunotherapy of Advanced Hepatobiliary Malignancy
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Deputy Director, Ruijin Hospital
Other Study IDs: RuijinH 2024-232
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-09

CONDITIONS: Hepatobiliary Malignancy
Keywords: 68Ga-grazytracer PET/CT; Immunotherapy; Advanced hepatobiliary malignancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosis of advanced hepatobiliary malignancies: Patients diagnosis of advanced hepatobiliary malignancies require immunotherapy or combination immunotherapy after evaluation according to clinical guidelines

SUMMARY:
This study aims to investigate the value of 68Ga-grazytracer in predicting the efficacy of immunotherapy for advanced hepatobiliary malignancies.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo a 68Ga-grazytracer PET/CT after 3 cycles of immunotherapy to evaluate response. The imaging response measurements will be compared with the histopathological or clinical assessment results as gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological and clinical diagnosis of advanced hepatobiliary malignancy requiring immunotherapy or combination immunotherapy after evaluation according to clinical guidelines
2. Signed and dated informed consent form
3. Commitment to comply with research procedures and co-operation in the implementation of the full research process
4. aged 18-75 years old
5. The patient is in good general condition with an expected survival of > 6 months

Exclusion Criteria:

1. Patients with serious illnesses that researchers consider unsuitable for participation in this clinical study. Such as severe heart and lung failure, severe bone marrow suppression, severe liver and kidney dysfunction, etc.
2. Intestinal perforation, complete intestinal obstruction
3. Uncontrolled diabetes patients or fasting blood glucose levels ≥11 mmol/L on the day of the trial
4. Pregnant women and women who may be pregnant, women who are breastfeeding.
5. Non-compliant person

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients at Ruijin Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation the responses to immunotherapy of advanced hepatobiliary malignancy | up to 9 weeks
  The value of 68Ga-grazytracer PET in monitoring responses to immunotherapy of advanced hepatobiliary malignancy
Standardized uptake value(SUV) | up to 9 weeks
  SUV of 68Ga-grazytracer uptake on PET/CT images for tumor lesions
Target-to-background ratio(TBR) | up to 9 weeks
  68Ga-grazytracer uptake ratio of tumor lesions to mediastinum and liver blood pool on PET/CT images.

SECONDARY OUTCOMES:
Progress free survival | 1 years
  Progress free survival
Overall survival | 1 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No